CLINICAL TRIAL: NCT03171064
Title: Sportivumab - Feasibility of Exercise as a Supportive Measure for Patients Undergoing Checkpoint-inhibitor Treatment
Brief Title: Exercise as a Supportive Measure for Patients Undergoing Checkpoint-inhibitor Treatment
Acronym: Sportivumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Department of Dermatology, Heidelberg University Hospital (Unknown)
Responsible Party: Principal Investigator, Joachim Wiskemann, Dr. Joachim Wiskemann, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Sportivumab/S-103/2017
Record Dates: First submitted 2017-05-24; First posted 2017-05-31 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: PD-1 Antibodies; Exercise; Melanoma
Keywords: Exercise; Cancer; Melanoma; Feasibility; PD-1 antibodies; Checkpoint inhibitors; Immune system
MeSH Terms: conditions — Motor Activity; Melanoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental intervention arm (EX) (Experimental): The supervised progressive endurance and resistance exercise program will be undertaken twice weekly in small groups and will be guided by an exercise physiotherapist over 12 weeks. All sessions will start with a warm-up passing over to the endurance training part and finish with a cool-down and will take approximately 60 minutes. The moderate-to-high-intensity endurance training will be performed at the beginning of each training session on a cycle ergometer for 20 min at 75 to 80 % of peak heart rate obtained from the baseline cardiorespiratory exercise test. This training intensity is within the range of intensities recommended by the American College of Sports Medicine (ACSM) exercise guidelines for cancer survivors. The moderate-to-high-intensity progressive resistance training regime (12 repetition maxima - 3 sets for each exercise) will include 6 exercises that target major upper and lower body muscle groups.
  Interventions: Behavioral: Resistance and Endurance Exercise
- Wait list - control group (UC) (No Intervention): Wait list control group will receive usual care. After primary endpoint assessment, UC patients will be offered to participate in the exercise interventions program.

INTERVENTIONS:
Behavioral: Resistance and Endurance Exercise — Machine-based, 2x/week endurance and resistance training for 12 weeks
  Arms: Experimental intervention arm (EX)

SUMMARY:
Checkpoint inhibitors like the PD-1 antibodies Pembrolizumab and Nivolumab represent standard of care for patients with metastasized melanoma. Numerous high quality studies demonstrate that endurance and resistance training in cancer patients is safe and elicits beneficial effects. However, there is no systematic experience with regard to exercise interventions in patients undergoing checkpoint inhibitor treatment. Therefore, the Sportivumab Study aimed to investigate safety, feasibility and effectivity of a 12 week combined resistance and endurance exercise intervention program during checkpoint inhibitor treatment. It is planned to enroll 40 patients. Participants will be randomized into an experimental and a wait-list control group (20 per group). The wait-list control group will receive the exercise intervention program after week 13 of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patients at age ≥ 18 years
* Diagnosed with melanoma stage (independent of stage)
* Assigned to receive an immunotherapeutic regimen (PD-1 antibody +/- Ipilimumab)
* Sufficient German language skills
* Willing to train at the exercise facilities twice per week and to take part in the scheduled testing at the National Center for Tumor Diseases
* Signed informed consent

Exclusion Criteria:

* Any physical or mental conditions that would hamper the performance of the training programs or the completion of the study procedures
* Engaging in systematic intense exercise training (at least 1h twice per week)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of the exercise intervention | During 12 week of the intervention
  Participants ability to fulfill the exercise prescription (measured by % of training frequency, intensity and duration as well as type of the exercise) during immune checkpoint inhibitor treatment with a PD-1 antibody +/- ipilimumab

SECONDARY OUTCOMES:
Quality of life | During 12 week of the intervention
  Quality of life (QoL) will be assessed with the validated 30-item self-assessment questionnaire of the European Organisation for Research and Treatment of Cancer (EORTC QLQ-C30, version 3.0). It includes five multi-item functional scales (physical, role, emotional, cognitive, and social function), three multi-item symptom scales (fatigue, pain, nausea/vomiting), and six single items assessing further symptoms (dyspnea, insomnia, appetite loss, constipation, diarrhea) and financial difficulties.
Fatigue | During 12 week of the intervention
  Fatigue will be assessed with the Multidimensional Fatigue Inventory (MFI) which is a 20-item, multidimensional self-assessment questionnaire that has been validated for a German-speaking population.It covers five different dimensions of fatigue (general fatigue, physical fatigue, reduced activity, reduced motivation, and mental fatigue).
Sleep Quality | During 12 week of the intervention
  Sleep quality and sleep problems will be assessed with the validated and frequently used Pittsburgh Sleep Quality Index (PSQI).
Depression | During 12 week of the intervention
  Depressive symptoms are assessed with the 20-item Center for Epidemiological Studies Depression Scale (CES-D).
Physical Activity Behavior | During 12 week of the intervention
  Physical activity (PA) behavior in the domains of commuting activity, leisure time activities such as cycling, walking, and sports, household and occupational activity will be assessed via a standardized and validated questionnaire, the Short QUestionnaire to ASsess Health-enhancing PA (SQUASH) which has the advantage that it is short and easy to complete.
Cardiopulmonary Fitness | During 12 week of the intervention
  Cardiopulmonary fitness will be measured by assessing maximal aerobic capacity (VO2peak) via a maximal incremental cycling test with a quasi-ramp protocol starting at 20 watts and increasing by 10 watts every minute until volitional exhaustion. To control for test validity gas exchange will be measured using a breath-by-breath gas analysis system which will be calibrated according to the instructions of the manufacturer before each test. To monitor patient safety, a 12-lead electrocardiogram (ECG) will be and blood pressure will be measured prior, during and after testing. The criteria for exhaustion will be fulfilled if two out of three of the following criteria are valid: (1) Borg scale > 16; (2) peak heart rate ± 10% of age-appropriate reference value and/or (3) respiratory exchange ratio (RER) > 1.1. Exercise will be terminated prematurely in the case of major ECG abnormalities, severe dyspnea or excessive blood pressure increase (≥250 mmHg systolic and/or ≥110 mmHg diastolic).
Muscle strength | During 12 week of the intervention
  Isometric (in four different joint angle positions) and isokinetic (at 60° angle speed) muscle capacity is measured with the Isomed 2000® diagnostic module (isokinetic evaluation and training machine). The protocol includes testing of representative muscles groups for upper (elbow flexors/extensors) and lower extremity (knee extensors/flexors)
Pain | During 12 week of the intervention
  The Brief Pain Inventory (BPI) is a 14-item questionnaire developed for use in patients with cancer that assesses worst pain, pain severity, and pain interference over the past week, reported on a scale of 0 to 10. Worst pain is categorized as mild (score of 3 to 4), moderate (score of 5 to 7), or severe pain (score of 8 to 10). Pain severity is measured as the average of responses to questions on worst pain, average pain, least pain, and pain right now. Pain interference is the average of seven interference items, such as walking, mood, and sleep.

CONTACTS AND LOCATIONS:
Locations (1):
- Heidelberg University Clinic, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Maybe pooling data with a comparable project in the united states